CLINICAL TRIAL: NCT03145558
Title: TATE Versus TACE, an Open-label Randomized Study Comparing TransArterial Tirapazamine Embolization Versus TransArterial ChemoEmbolization in Intermediate Stage Hepatocellular Carcinoma
Brief Title: TATE Versus TACE in Intermediate Stage HCC
Acronym: TATE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Landscape changed and the study population is no longer suitable for the study treatment.
Sponsor: Teclison Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LT-006
Record Dates: First submitted 2017-05-03; First posted 2017-05-09 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Tirapazamine, embolization, TACE, Hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Tirapazamine; Doxorubicin

STUDY DESIGN:
Intervention Model Description: 1:1 randomization, open label with central radiological review
Who Masked: Outcomes Assessor
Masking Description: Central radiology reviewers are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Trans-Arterial Tirapazamine Embolization (TATE) (Experimental): Patients will receive a fixed dose of Tirapazamine combined with embolization using Lipiodol and Gelfoam.
  Interventions: Drug: Tirapazamine
- Trans-Arterial ChemoEmbolization (TACE) (Active Comparator): Patients will receive a mixture of doxorubicin and Lipiodol into the tumor feeding artery followed by injection of Gelfoam to induce embolization per standard procedure.
  Interventions: Drug: Doxorubicin

INTERVENTIONS:
Drug: Tirapazamine — Replacing the standard chemotherapy agent doxorubicin used in TACE with tirapazamine
  Arms: Trans-Arterial Tirapazamine Embolization (TATE)
Drug: Doxorubicin — Standard of care for TACE
  Arms: Trans-Arterial ChemoEmbolization (TACE)

SUMMARY:
An open label randomized study to compare TATE versus TACE in patients with intermediate stage Hepatocellular carcinoma who are not suitable for surgical resection or radiofrequency ablation. The primary endpoint is Progression Free Survival. Secondary endpoints including CR rate, Time to embolization failure, Duration of CR, OS, ORR, local control rate, time to local recurrence and duration to local recurrence. The study treatment is to compare Tirapazamine versus doxorubicin when combined with trans-arterial embolization. Study plans to enroll 134 patients in 1:1 randomization for TATE or TACE. MRI will be used to assess efficacy using a central radiological review for the final analysis.

DETAILED DESCRIPTION:
Trans-arterial chemoembolization (TACE) is a standard care of intermediate stage Hepatocellular carcinoma (HCC) for 40 years without much improvement in efficacy. The key reason for lack of progress is that chemotherapy agents are not effective in hypoxia and cancer stem cells are induced under hypoxia. Tirapazamine, a hypoxia activated agent, can potential solve these two problems. This open label randomized trial will be conducted in HCC patients who are in intermediate stage and naive to embolization, Child Pugh up to B7 and with normal organ functions. Patients will be randomized 1:1 to receive TATE (trans-arterial tirapazamine embolization) or conventional TACE. The goal of treatment aims to achieve CR by mRECIST for every patient. If there is evidence of viable lesion, patients should be treated again. All patients are followed by contrast MRI scans every 2 months in the first year and every 3 months afterwards until patients have evidence of progression and no longer considered suitable for TATE/TACE. Survival will be followed for 3 years. Total sample size will be 134 patients with the total study duration for 3 years.

ELIGIBILITY:
1. Confirmed diagnosis of HCC by imaging criteria per American Association for the Study of Liver Diseases (AASLD) criteria.
2. Patients with single or multiple HCC who are unsuitable for surgical resection or RFA, but suitable for embolization.
3. ECOG score 0-1. Child-Pugh score up to B7.
4. Patients should have measurable tumor lesion(s) by contrast MRI.
5. Patients have adequate normal organ function and suitable laboratory criteria.
6. Men and women of child-bearing age need to commit to using two levels of contraception simultaneously to avoid pregnancy.

Exclusion Criteria:

1. Patients who have had a liver transplantation.
2. Patients who have uncontrolled major medical problems such as cardiac, pulmonary (COPD requiring constant oxygen), renal (creatinine over 2.0) diseases, active infectious diseases (except chronic Hepatitis B or C), or non-healing ulceration.
3. Patients who have any clinical evidence of hypoxia with O2 saturation less than 92% on room air.
4. Patients with evidence of arterial insufficiency or microangiopathy in any organ due to any reason, which could lead to distal extremity hypoxia, as evidenced by any gangrenous change in distal limbs or requiring resection for this reason.
5. Patients with poorly controlled HBV infection.
6. Patients on interferon treatment need to have at least 2-week washout period from Day 1.
7. Patients with major gastrointestinal bleeding in the prior 2 months of enrollment or known diagnosis of cancer other than HCC.
8. Pregnant or lactating women.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | within 2 years
  mRECIST criteria

SECONDARY OUTCOMES:
Overall survival | 3 years
  From randomization to death
Complete Response rate | 2 years
  CR rate based on mRECIST criteria
Time to Embolization Failure | 1 year
  From randomization to stage progression
Duration of CR | 1 year
  From randomization to recurrence in those patients who achieved CR

OTHER OUTCOMES:
Local recurrence rate | 1 year
  Recurrence rate in the embolized lesion
Time to local recurrence | 2 years
  From randomization to local recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Abi-Jaoudeh, Study Chair — University of California, Irvine
Locations (3):
- United States (3):
  - University of California, Irvine, Irvine, California
  - Oregon Health Science University, Portland, Oregon
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No